CLINICAL TRIAL: NCT04158063
Title: Cognitive-motor Interference in Persons With MS: Dual Task Assessment and Training - A Multi-center Study
Brief Title: Cognitive-motor Interference in Persons With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other); AZ Klina (Other); Centre Hospitalier Universitaire de Liege (Other); Masku Neurological Rehabilitation Centre (Unknown); Tel Aviv University (Other); Sheba Medical Center (Other Government); AISM Rehabilitation Service of Genoa (Unknown)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCS-IV-CMI&DTT-01
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: knows what kind of training, but not whether the trainings-group is the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Training (DTT) (Experimental)
  Interventions: Behavioral: Dual Task Training
- Single Mobility Training (SMT) (Active Comparator)
  Interventions: Other: Single Mobility Training

INTERVENTIONS:
Behavioral: Dual Task Training — In total 12 Dual Task conditions will be performed in which 3 cognitive tasks are combined with 4 motor tasks:
  Cognitive tasks:
  * Titrated digit span backwards
  * Auditory vigilance with alphabets
  * Subtracting by 7
  Motor tasks:
  * Walking at self-selected speed
  * Walking while carrying a cup of water
  * Walking while stepping over obstacles
  * Walking crisscross
  Arms: Dual Task Training (DTT)
Other: Single Mobility Training — standard routine training
  Arms: Single Mobility Training (SMT)

SUMMARY:
Dual tasking such as walking while talking on the phone or while remembering a shopping list is very frequently required in everyday life. Cognitive-motor interference occurs when the performance capacity of a motor or cognitive task decreases when both are performed simultaneously (dual task) compared to single task execution being the so-called dual task cost (DTC). Over the past five years, in MS, (pilot) studies have been conducted in order to investigate the presence and magnitude of the CMI during walking. It was shown that, even in the early stages of the disease, when walking speed is not affected as a single motor task, pwMS slow down more than healthy controls when performing DT walking. Studies have not yet investigated the impact of the complexity of the motor task, on the DTC. Across studies, many different types of cognitive distractors were applied without any documentation of psychometric properties, such as test-retest reliability, making it not yet suited as experimental outcome measure. Results have also focused on the effects of DT on walking performance, while the performance of the cognitive task was rarely assessed. Also, the majority of studies did not document the cognitive function level of pwMS or even excluded patients with cognitive deficits. As such, the relation between cognitive deficits and dual task (cognitive-motor) performance is unclear.

Motor and cognitive impairment are currently also treated separately whereas real life performance very often requiring an integrated motor and cognitive function. So far, no studies in MS have investigated the effects of physical or cognitive exercises on DT performances, or investigated effects of integrated cognitive-motor dual task training (DTT). In elderly and other neurological conditions, superior effects of dual task training (DTT) on gait training have been suggested, but the evidence is not robust yet. All these studies suggest the feasibility of DTT on gait improvement and fall risk reduction, but further insights on factors identifying responders, and differential effect of cognitive distractors needs further elucidation.

This research consist of two parts that aim to investigate:

Part 1: Assessment

1. the magnitude of the dual task cost according to different types of cognitive distractors (information processing, memory, attention, etc.),
2. its reliability as experimental outcome measure and
3. its association with factors as severity of cognitive or motor dysfunction, quality of life and fatigue.

Part 2: Intervention

1. the effectiveness of cognitive-motor DT-based training programs compared to single modality training, on DT and ST performances (cognition and mobility)
2. whether dual task learning effects transfer to improvements in daily life and are sustained for 4 weeks without training
3. which patient profiles benefit most from the integrated cognitive-motor training
4. feasibility and usefulness of an adaptive, interactive ICT-guided DTT system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to McDonald criteria
* EDSS ≥2 and ≤ 6
* No relapse within the last 30 days
* No changes in disease modifying treatment and no corticoid-therapy within the last 50 days
* All types of MS
* Minimal cognitive functioning (MMSE≥26)
* Presence of dual task interference (dual task screening list ≥1)

Exclusion Criteria:

* Other medical conditions interfering with mobility
* Other neurological diagnoses
* MS-like syndroms such as neruomyelitis optica
* Not able to understand and execute simple instructions
* Problems (even after adjustment with hearing aids or glasses) with hearing or vision interfering with the assessment or training.
* Ongoing dual task training or other interfering physical therapy or cognitive training/neuropsychological rehabilitation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Digit Span - Walk - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 - 5 4 1
Digit Span - Walk - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 - 5 4 1
Digit Span - Walk - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 - 5 4 1
Subtraction - Walk - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.)
Subtraction - Walk - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.)
Subtraction - Walk - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.)
Vigilance - Walk - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Walk - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Walk - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Digit Span - Cup - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Cup - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Cup - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Subtraction - Cup - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Subtraction - Cup - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 ->145 - 138 - 131, etc.).
Subtraction - Cup - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Vigilance - Cup - Dual Task Cost (%) | baseline
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard
Vigilance - Cup - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard
Vigilance - Cup - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed with a cup filled with water in the hand on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard
Digit Span - Obstacles - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Obstacles - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Obstacles - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Subtraction - Obstacles - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Subtraction - Obstacles - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 ->145 - 138 - 131, etc.).
Subtraction - Obstacles - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Vigilance - Obstacles - Dual Task Cost (%) | Baseline
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Obstacles - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Obstacles - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked at self-selected speed while stepping over obstacles placed every 3 meters on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Digit Span - Crisscross - Dual Task Cost (%) | baseline
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Crisscross - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Digit Span - Crisscross - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the titrated digit span backwards. The titrated digit span backward is a task in which the participant hears a string of numbers that they have to repeat in reverse order (f.e. 1 4 5 -> 5 4 1).
Subtraction - Crisscross - Dual Task Cost (%) | Baseline
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Subtraction - Crisscross - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Subtraction - Crisscross - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the serial subtraction with sevens task. The serial subtraction with sevens task is a task in which the participant was given a starting number of 3 digits (e.g. 152) from which they had to continuously subtract sevens (f.e. 152 -> 145 - 138 - 131, etc.).
Vigilance - Crisscross - Dual Task Cost (%) | Baseline
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Crisscross - Dual Task Cost (%) | Week 9 (post-measure)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.
Vigilance - Crisscross - Dual Task Cost (%) | week 13 (4-week follow-up)
  persons walked crisscross from cone to cone every 2m with 80cm fixed width in between at self-selected speed on a 30-meter walkway for 1 minute, while performing the vigilance task. The vigilance task is a task in which the participants listened to letters of the alphabet and had to say aloud 'yes' every time they heard 1 of the 2 target letters (e.g. 'L' or 'R') and were asked not to respond when another letter was heard.

SECONDARY OUTCOMES:
Brief Repeatable Battery of Neuropsychological Tests | baseline
  This battery consists of six tests in different cognitive domains: 1) the Selective Reminding test, 2) the 10/36 spatial recall test, 3) the symbol digit modalities test, 4) the Paced auditory serial addition test with 3 seconds, 5) the Paced auditory serial addition test with 2 seconds and 6) the word list generation.
Part of Brief Repeatable Battery of Neuropsychological Tests | Week 9 (post-measure)
  The symbol digit modalities test, the Paced auditory serial addition test with 3 seconds and the Paced auditory serial addition test with 2 seconds were assessed.
Part of Brief Repeatable Battery of Neuropsychological Tests | week 13 (4-week follow-up)
  The symbol digit modalities test, the Paced auditory serial addition test with 3 seconds and the Paced auditory serial addition test with 2 seconds were assessed.
Multiple Sclerosis Impact Scale-29 (MSIS-29) | baseline
  Questionnaire to record participants' perceived impact of MS on day-to-day life.
  a 29-item self-report measure comprised of 20 items associated with a physical scale and 9 items associated with a psychological scale.1 Items question patients (or their proxies) about the impact of multiple sclerosis (MS) on day-today life in the last 2 weeks. All items have 5 response options from 1 (not at all) to 5 (extremely). Each of the 2 scales are scored by summing the responses across items, then converting to a 0 to 100 scale, where 100 indicates greater impact of disease on daily function (worse health).
Multiple Sclerosis Impact Scale-29 (MSIS-29) | Week 9 (post-measure)
  Questionnaire to record participants' perceived impact of MS on day-to-day life.
  a 29-item self-report measure comprised of 20 items associated with a physical scale and 9 items associated with a psychological scale.1 Items question patients (or their proxies) about the impact of multiple sclerosis (MS) on day-today life in the last 2 weeks. All items have 5 response options from 1 (not at all) to 5 (extremely). Each of the 2 scales are scored by summing the responses across items, then converting to a 0 to 100 scale, where 100 indicates greater impact of disease on daily function (worse health).
Multiple Sclerosis Impact Scale-29 (MSIS-29) | week 13 (4-week follow-up)
  Questionnaire to record participants' perceived impact of MS on day-to-day life.
  a 29-item self-report measure comprised of 20 items associated with a physical scale and 9 items associated with a psychological scale.1 Items question patients (or their proxies) about the impact of multiple sclerosis (MS) on day-today life in the last 2 weeks. All items have 5 response options from 1 (not at all) to 5 (extremely). Each of the 2 scales are scored by summing the responses across items, then converting to a 0 to 100 scale, where 100 indicates greater impact of disease on daily function (worse health).
Modified Fatigue Impact Scale (MFIS) | baseline
  This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial. The MFIS is a 21-item questionaire, scale 0 (never)-4 (always), scale range 0-40
Modified Fatigue Impact Scale (MFIS) | Week 9 (post-measure)
  This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial. The MFIS is a 21-item questionaire, scale 0 (never)-4 (always), scale range 0-40
Modified Fatigue Impact Scale (MFIS) | week 13 (4-week follow-up)
  This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial. The MFIS is a 21-item questionaire, scale 0 (never)-4 (always), scale range 0-40
Dual Task Questionnaire | Baseline
  Questionnaire to record participants' perception of dual task problems in daily life.
Dual Task Questionnaire | Week 9 (post-measure)
  Questionnaire to record participants' perception of dual task problems in daily life.
Dual Task Questionnaire | week 13 (4-week follow-up)
  Questionnaire to record participants' perception of dual task problems in daily life.
Timed 25 Foot-walk test (T25FW) | baseline
  test of motor function in which participants walk 25-foot.
Timed 25 Foot-walk test (T25FW) | Week 9 (post-measure)
  test of motor function in which participants walk 25-foot.
Timed 25 Foot-walk test (T25FW) | week 13 (4-week follow-up)
  test of motor function in which participants walk 25-foot.
Timed-up-and-go test (TUG) | baseline
  test of walking and balance in which participants stand up from a chair, walk, turn and sit down again.
Timed-up-and-go test (TUG) | Week 9 (post-measure)
  test of walking and balance in which participants stand up from a chair, walk, turn and sit down again.
Timed-up-and-go test (TUG) | week 13 (4-week follow-up)
  test of walking and balance in which participants stand up from a chair, walk, turn and sit down again.
Dynamic Gait Index (DGI) | Baseline
  test in which assessor scores gait performance of the participant.
Dynamic Gait Index (DGI) | Week 9 (post-measure)
  test in which assessor scores gait performance of the participant.
Dynamic Gait Index (DGI) | week 13 (4-week follow-up)
  test in which assessor scores gait performance of the participant.
2-minute walking test (2MWT) | baseline
  test of walking in which participants walk for 2 minutes
2-minute walking test (2MWT) | Week 9 (post-measure)
  test of walking in which participants walk for 2 minutes
2-minute walking test (2MWT) | week 13 (4-week follow-up)
  test of walking in which participants walk for 2 minutes
Multiple sclerosis walking scale-12 (MSWS-12) | baseline
  questionnaire to measure perception of limitations in walking ability caused by MS.
Multiple sclerosis walking scale-12 (MSWS-12) | Week 9 (post-measure)
  questionnaire to measure perception of limitations in walking ability caused by MS.
Multiple sclerosis walking scale-12 (MSWS-12) | week 13 (4-week follow-up)
  questionnaire to measure perception of limitations in walking ability caused by MS.
Falls efficacy scale (FES-I) | baseline
  uestionnaire to measure concerns about the possibility of falling.
Falls efficacy scale (FES-I) | Week 9 (post-measure)
  uestionnaire to measure concerns about the possibility of falling.
Falls efficacy scale (FES-I) | week 13 (4-week follow-up)
  uestionnaire to measure concerns about the possibility of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Ilse Baert, drs., Study Chair — Hasselt University; Renee Veldkamp, drs., Study Chair — Hasselt University
Locations (1):
- Revalidatie & MS Centrum Overpelt, Overpelt, Belgium